CLINICAL TRIAL: NCT03906487
Title: Self Defining Memories in Women Victims of Intimate Partner Violence: a Pilot Study.
Brief Title: Self Defining Memories in Women Victims of Intimate Partner Violence.
Acronym: SOI-MEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/19/0051
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Domestic Violence
Keywords: Intimate partner violence; Self defining memories

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intimate partner violence (Experimental): The women in this arm must have suffered at least two physical aggressions. They will be recruited in the study as part of their coming to the consultation of intentional injury of the medico-legal unit of the University Hospital Toulouse.
  Interventions: Behavioral: Assessment measures MINI, PCL5 and BDI-II and definition of 5 SDM
- Control group (Active Comparator): The women in this group are women who have never experienced domestic violence or have experienced a potentially traumatic event. These women will be recruited by a call for volunteers.
  Interventions: Behavioral: Assessment measures MINI and definition of 5 SDM

INTERVENTIONS:
Behavioral: Assessment measures MINI, PCL5 and BDI-II and definition of 5 SDM — This group will have two visits:
  * the first to verify inclusion criteria and assessed psychotraumatic and depressive symptoms by completing assessment measures called MINI, PCL-5, BDI-II ;
  * the last to characterize the SDM by defining 5 personal memories
  Arms: Intimate partner violence
Behavioral: Assessment measures MINI and definition of 5 SDM — This group will have two visits:
  * the first to verify inclusion criteria and assessed psychotraumatic and depressive symptoms by completing MINI questionary;
  * the last to characterize the SDM by and defining 5 personal memories
  Arms: Control group

SUMMARY:
A recent report by the World Health Organization demonstrated that 30 % of women worldwide have been victims of intimate-partner violence (IPV). IPV is a public health problem thus it seems important to propose relevant care. It is difficult to carry out an effective therapy. Psychological care is based on cognitive abilities but these women have cognitive impairment. Few studies investigated their cognitive dysfunction. Investigators suggest in this study an exploration of the Self Defining Memories (SDM) which can highlight the loss of identity of these women and a new target of therapy.

DETAILED DESCRIPTION:
Intimate partner violence among women is associated to identity problems. Indeed, the victims have a poor self esteem and difficulties to express their own wishes. In this study investigators suggest an analysis of a type of memory, that is known to be essential, to profile an identity functioning: self-defining memories. To date, no study has explored SDM in women with IPV. The characteristics of the SDM in women victims of IPV will be compared to a group of women who has never been diagnosed in this situation. Those memories could be used in therapy. A French adaptation of the questionnaire proposed by Singer & Moffitt (1992) will be used (Berna et al., 2011a, 2011b) for the assessment of SDM.

Four elements will be study: specificity, meaning, content, affect.

The two groups will have two visits:

* the first to verify inclusion criteria and assessed psychotraumatic and depressive symptoms;
* the last to characterize the SDM.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* French mother tongue.
* Informed consent.
* Affiliated to social security

For women who are victims of IPV only:

* Having at least two physical aggressions
* To meet criterion A of the diagnosis of PTSD according to the Diagnostic and Statistical Manual of Mental Disorders DSM (DSM-5) (evaluated using the Mini International Neuropsychiatric Interview, MINI)

For women of the control group only:

- None a victim of IPV

Exclusion Criteria:

For all participants:

* Neurological pathology, brain damage.
* History of head trauma with loss of consciousness.
* Severe, progressive somatic pathology
* Psychotherapy in progress
* Taking psychotropic drugs or beta-blockers (because of their potential impact on memory capacity)
* Pregnant or lactating women
* Under a legal regime for the protection of adults

For women who are victims of IPV only:

* Antecedent or presence of PTSD other than that related to IPV
* History or presence of progressive mental disorders (Axis I DSM-5 - evaluated using Mini International Neuropsychiatric Interview, MINI)

For women of the control group only:

History or presence of progressive mental disorders including PTSD (Axis I DSM-5 - evaluated using Mini International Neuropsychiatric Interview, MINI)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Description of five Self Defining Memories. | 7 to 10 days after inclusion visit
  These memories are declined in four dimensions: specificity, content, meaning and emotional valence. Investigator will get a proportion of memories which are specific, which are negative, positive or neutral, which have an integrative meaning and which are associated to violence for IPV victims. The results of Self Defining Memories will be compared between a group of IPV victims and a control group.

SECONDARY OUTCOMES:
Proportions of SDM whose content is associated with discomfort in IPV victims compared to those of control. | 7 to 10 days after inclusion visit
Proportions of SDM whose emotional valence is associated with a feeling of redemption or contamination in IPV victims compared to those of control. | 7 to 10 days after inclusion visit
Relationships between the 4 dimensions of SDM and psychotraumatic symptoms in IPV victims. | 7 to 10 days after inclusion visit
  These symptoms will be measured via the Posttraumatic Stress Disorder Checklist (PCL-5 scale).This is a self-questionnaire to assess the main symptoms of Post traumatic stress disorder. It has 20 items that evaluate the intensity and frequency of symptoms in the previous month using scores from 1 to 4.The higher the score, the more important the trauma.
Relationships between the 4 dimensions of SDM and depressive symptoms in IPV victims. | 7 to 10 days after inclusion visit
  These symptoms will be measured via the Beck Depressin Inventory (BDI) scale: this is a self-questionnaire to assess the severity of depressive symptoms using 21 items. Once the test is completed, a score is made by decounting, then compared according to the score, thus determining the severity of the depression:
  0 - 9: indicates a minor depression 10 - 18: indicates slight depression 19 - 29: indicates moderate depression 30 - 63: indicates severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Damien PIERRE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France